CLINICAL TRIAL: NCT06904092
Title: Efficacy and Mechanisms of Transcranial Ultrasound Stimulation (TUS) on Cognitive Deficits in Schizophrenia：based on the Hippocampal-Prefrontal Circuit
Brief Title: Efficacy and Mechanisms of TUS on Cognitive Deficits in Schizophrenia: Based on the Hippocampal-Prefrontal Circuit
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 82371504
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Deficit in Schizophrenia
Keywords: Schizophrenia; Cognitive Deficit; Transcranial Ultrasound Stimulation; Hippocampus- Prefrontal Circuit
MeSH Terms: conditions — Schizophrenia; Cognition Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- single target group : left DLPFC (Active Comparator): 35 eligible patients will be treated with active TUS for 4 weeks on the left DLPFC
  Interventions: Device: Transcranial ultrasound stimulation
- single target group : left hippocampus (Active Comparator): 35 eligible patients will be treated with active TUS for 4 weeks on the left hippocampus
  Interventions: Device: Transcranial ultrasound stimulation
- both-target group : left DLPFC and left hippocampus (Active Comparator): 35 eligible patients will be treated with active TUS for 4 weeks on the left DLPFC and left hippocampus
  Interventions: Device: Transcranial ultrasound stimulation

INTERVENTIONS:
Device: Transcranial ultrasound stimulation — The TUS was administered using Transcranial Ultrasound Stimulator UNS-III (model UNS-III), which has passed the safety test for medical electrical equipment (GB9706.1-2007). Transcranial ultrasound stimulation on the target. Duration:20 days (workdays for four consecutive weeks).

SUMMARY:
Cognitive deficit is a core symptom of schizophrenia related to poorer functional outcome. Prior studies indicated that abnormalities in the hippocampus-prefrontal circuit and glutamate/GABA imbalances may lead to cognitive deficits. Based on the current background and our previous studies, it has been proved that TUS can modulate neural excitability and plasticity in the hippocampus. In this double-blind, randomized study, the efficacy of different treatment options and mechanisms of TUS on cognitive deficits will be investigated.

DETAILED DESCRIPTION:
Cognitive deficit is a core symptom of schizophrenia related to poorer functional outcome which remains largely treatment refractory. Prior studies indicated that abnormalities in the hippocampus-prefrontal circuit and glutamate/GABA imbalances may be the root causes of cognitive deficits. Transcranial ultrasound stimulation (TUS), an emerging non-invasive neuromodulation technique with deep penetration ability, can modulate neural excitability and plasticity in the hippocampus. This is a 4-week double-blind randomized trial of TUS for cognitive deficits in schizophrenia, with either left hippocampus or left dorsolateral prefrontal cortex (DLPFC) or both targeted. This study aims to determine the efficacy of TUS and to reveal its underlying neural mechanism, especially with the hippocampus-prefrontal circuit, by means of TUS, as to assess cortical inhibition and excitability, EEG source imaging, and multi-model MRI. Neuropsychological assessments will also be conducted to develop the optimized treatment strategy. The study points to a novel and promising therapeutic neuromodulation approach that may improve the functional outcome of schizophrenia, which has been the main cause of mental disability.

ELIGIBILITY:
Inclusion Criteria:

* Meet the DSM-5 diagnostic criteria for schizophrenia ;
* Age18-50, right-handed, Han nationality;
* Presence of cognitive deficit: defined as d' value <0.5 in associative memory test;
* Be in a stable condition, received second-generation antipsychotics for at least 4 weeks or more;
* Written informed consent;

Exclusion Criteria:

* Current or past neurological illness, severe physical diseases, substance abuse or alcohol dependence, mental retardation, pregnancy or lactation;
* Uncooperative or risky patients with high excitement, stupor, disorder of words and deeds, negative suicide, etc.;
* History of MECT or other physical therapy within 6 months;
* History of epilepsy, or epileptic waves on the baseline EEG;
* Ruled out share antiepileptic drugs (carbamazepine, valproic acid salt) or larger doses of benzodiazepine drugs (diazepam > 10mg/day, clonazepam > 2mg/day etc.), if necessary, remain unchanged during the course of treatment;
* Contraindications to TUS and MRI are present.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in associative memory test score | baseline, 4 weeks and 8 weeks
  Change from baseline in the associative memory test score at 4 weeks and 8 weeks.

SECONDARY OUTCOMES:
Change of information processing speed and attention/vigilance | baseline, 4 weeks and 8 weeks
  Change from baseline in 4 MCCB subtests score at 4 weeks and 8 weeks.
Change of working memory | baseline, 4 weeks and 8 weeks
  Change from baseline in N-back task at 4 weeks and 8 weeks. The outcome measures include accuracy, D-prime value, and reaction time.
Change from baseline in Positive and Negative Syndrome Scale(PANSS) | baseline, 4 weeks and 8 weeks
  Change from baseline in Positive and Negative Syndrome Scale(PANSS) at 4 weeks and 8 weeks. The minimum to maximum value is 30-210. Lower scores mean a better outcome.
Change of CGI score | baseline, 4 weeks and 8 weeks
  Change from baseline in Clinical Global Impression (CGI) at 4 weeks and 8 weeks.
Change from baseline in UCSD Performance-based Skills Assessment-Brief (UPSA-B) | baseline, 4 weeks and 8 weeks
  Change from baseline in UCSD Performance-based Skills Assessment-Brief (UPSA-B) at 4 weeks and 8 weeks.
Change of Multi-modal Brain Neuroimaging in structure | baseline and 4 weeks
  Brain structure data will be acquired.
Change of Multi-modal Brain Neuroimaging in resting- state fMRI | baseline and 4 weeks
  Resting-state fMRI data will be acquired.
Change of Multi-modal Brain Neuroimaging in 1H-MRS | baseline and 4 weeks
  1H-MRS data will be acquired.
Change of TEPs | baseline and 4 weeks
  TMS-evoked potentials (TEPs) from target regions will be measured in participants at baseline, after a single TUS intervention, and at 4 weeks. The study aimed to clarify the effects of TUS treatment on the components of TEPs in individuals with schizophrenia, as well as the association between changes in TEP components and cognitive deficits.
Change of 64 channels EEG | baseline and 4 weeks
  64 channels EEG data will be acquired.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No